CLINICAL TRIAL: NCT00691665
Title: A Double-masked, Randomized, Parallel Group, Comparison of Olopatadine 0.6% and Fluticasone Proprionate 50mcg Nasal Sprays in a Two Week Seasonal Allergic Rhinitis Trial
Brief Title: Comparison of Olopatadine 0.6% and Fluticasone Proprionate 50mcg Nasal Sprays in a Two Week Seasonal Allergic Rhinitis Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Dr. Michael Edwards, PhD, Alcon Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMA-08-06
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinitis; Seasonal Allergic Rhinitis; allergies
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olopatadine HCL Nasal Spray, 0.6% (Experimental): Olopatadine HCL Nasal Spray, 0.6% 2 sprays per nostril twice daily
  Interventions: Drug: Olopatadine HCL Nasal Spray, 0.6%
- Fluticasone Propionate Nasal Spray, 50 mcg (Active Comparator): Fluticasone Propionate Nasal Spray, 50 mcg 2 sprays per nostril once daily
  Interventions: Drug: Fluticasone Propionate Nasal Spray, 50 mcg

INTERVENTIONS:
Drug: Olopatadine HCL Nasal Spray, 0.6% — Olopatadine HCL Nasal Spray, 0.6% 2 sprays per nostril twice daily
  Arms: Olopatadine HCL Nasal Spray, 0.6%
Drug: Fluticasone Propionate Nasal Spray, 50 mcg — Fluticasone Propionate Nasal Spray, 50 mcg 2 sprays per nostril once daily
  Arms: Fluticasone Propionate Nasal Spray, 50 mcg

SUMMARY:
Comparison of two nasal sprays for the treatment of seasonal allergic rhinitis

ELIGIBILITY:
Inclusion:

* A history of spring/summer seasonal allergies.
* Positive skin prick test for the currently prevalent allergen of the area.
* Confirmed absence of significant anatomic abnormalities, infection, bleeding, and mucosal ulcerations on nasal examination prior to administration of test article.
* For pre-menopausal females, a negative pregnancy test prior to entry into the study, and, if sexually active, agreement to use adequate birth control methods throughout the study.

Exclusion:

* History of chronic sinusitis.
* Asthma, with the exception of intermittent asthma.
* Smokers.
* Known non-responders to antihistamines.
* Chronic or intermittent use of inhaled, oral, intramuscular, intravenous or dermal potent or super-potent topical corticosteroids.
* Chronic use of long acting antihistamines.
* Upper or lower respiratory infection within 14 days of Visit 1. Diagnosis of acute sinusitis within 30 days of Visit 1.
* Relatives of study site staff or other individuals who had access to the clinical study protocol.
* Participation in any other investigational study within 30 days before entry into this study or concomitantly with this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sacramento, CA, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred from May 14, 2008 - July 31, 2008.
Period: Overall Study
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 2 | 10
  Between 18 and 65 years | 55 | 63 | 118
  >=65 years | 2 | 0 | 2
Gender [Number; unit: participants] — Gender information was not collected for 3 patients at baseline.
  participants
    Female | 34 | 30 | 64
    Male | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Reflective Total Nasal Symptom Score (rTNSS) From Baseline
Description: Responses to patient-completed diaries for reflective Total Nasal Symptom Scores (rTNSS). TNSS is composed of 4 individual assessments, which included runny nose, itchy nose, stuffy nose, and sneezing; each of the 4 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 4 assessments are then added together for a composite score (TNSS score), the maximum of which could be 12. Reflective scores were assessed from the hour since the last dose of study medication.
Time Frame: 14 Days minus baseline
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Number analyzed (Participants) | 65 | 65
Percent change | -45.37 (31.77) | -47.35 (32.83)

2. Primary Outcome: Mean Percent Change in Instantaneous Total Nasal Symptom Score (iTNSS) From Baseline
Description: Responses to patient-completed diaries for instantaneous Total Nasal Symptom Scores (iTNSS). TNSS is composed of 4 individual assessments, which included runny nose, itchy nose, stuffy nose, and sneezing; each of the 4 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 4 assessments are then added together for a composite score (TNSS score), the maximum of which could be 12. Instantaneous scores were assessed at the time of daily dosing.
Time Frame: 14 days minus baseline
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Number analyzed (Participants) | 65 | 65
Percent change | -45.26 (27.93) | -48.8 (30.10)

3. Primary Outcome: Mean Percent Change in Reflective Total Ocular Symptom Scores (rTOSS) From Baseline
Description: Responses to patient-completed diaries for reflective Total Ocular Symptom Scores (rTOSS). TOSS is composed of 3 individual assessments of ocular symptoms (itching/burning, tearing/watering, redness) each of the 3 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 3 assessments are then added together for a composite score (TOSS score), the maximum of which could be 9. Reflective scores were assessed from the hour since the last dose of study medication.
Time Frame: 14 Days minus baseline
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Number analyzed (Participants) | 65 | 65
Percent change | -38.52 (59.80) | -40.59 (55.66)

4. Primary Outcome: Mean Percent Change in Instantaneous Total Ocular Symptom Scores (iTOSS) From Baseline
Description: Responses to patient-completed diaries for instantaneous Total Ocular Symptom Scores (iTOSS). TOSS is composed of 3 individual assessments of ocular symptoms (itching/burning, tearing/watering, redness) each of the 3 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 3 assessments are then added together for a composite score (TOSS score), the maximum of which could be 9. Instantaneous scores were assessed at the time of daily dosing.
Time Frame: 14 Days minus baseline
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Number analyzed (Participants) | 65 | 65
Percent change | -36.54 (60.26) | -41.63 (50.46)

ADVERSE EVENTS:
Arm/Group | Olopatadine HCL Nasal Spray, 0.6% | Fluticasone Propionate Nasal Spray, 50 Mcg
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No